CLINICAL TRIAL: NCT05378438
Title: Impact of Microbe Literacy Initiative on Improved Vaccine Uptake in Peri-urban Slum Areas in Kathmandu, Nepal: A Community Based Cluster Randomized Controlled Trial
Brief Title: Impact of Microbe Literacy Initiative on Improved Vaccine Uptake in Peri-urban Slum Areas in Kathmandu, Nepal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nepal Health Research Council (Other Government)
Collaborators: Microbe Literacy Initiative (Unknown); Partnership for Sustainable Development Nepal (PSDNepal) (Unknown)
Responsible Party: Principal Investigator, Dr. Pradip Gyanwali,MD, Executive Chief, Nepal Health Research Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 39/2022
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Vaccine Acceptance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants allocated in this arm will be approached for a workshop related to microbe literacy. Using a microscope, live demonstration of the biological samples brought by the participants will be carried out by the team of researchers. Participants will be assisted to place biological materials under the microscope, manipulate the slides and discover the profusion of microbial life from the immediate environment. The session will be followed by question and answer round related to concurrent hygiene practices and basic sanitation to prevent infections including vaccines.
  Interventions: Other: Microbe literacy Program in the form of workshop
- Control arm (No Intervention): Participants in this arm will be consented for the study and baseline data collection will be made but there will not be any intervention. Data will be collected for baseline as well as post interventional vaccination status among the studied population.

INTERVENTIONS:
Other: Microbe literacy Program in the form of workshop — Two to Three hours of workshop on microbe literacy will be conducted as an intervention. Workshop includes discussion on various common microorganisms causing diseases, their sources, relationship with surroundings and management. Prime focus of the session will be on management via treatments and risk reduction via vaccination.
  Arms: Intervention Arm

SUMMARY:
This study is designed to assess the impact of the first introduction of microscope-based health education on people's attitude and practice towards disease prevention in Nepal, measured by vaccine acceptance rate. Such health education has an important role to play in communities where vaccine acceptance is low.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 years or older who are resident of the study target area
* People who stayed at least for 6 months on the area of study
* People who agrees with the procedure of study and follow ups visits
* People who provide consent for their participation will be recruited in the study.

Exclusion Criteria:

* People under 18 years of age will not be enrolled into study due to their limitation of understanding and implementation of the content of workshop given as intervention.
* People who do not wish to participate in the trial
* Those with currently ongoing court hearing and deprive of freedom will not be enrolled for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1252 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-04-17 (Estimated)

PRIMARY OUTCOMES:
Differential vaccine acceptance rates between intervention and control group | Within 3 months of intervention
  Data will be collected for baseline as well as post intervention after 3 months of workshop. For both the intervention and control group, number of vaccinated among the participants for provided COVID-19 vaccine and Typhoid vaccine will be made. Comparative analysis will be made in both the study groups before and after the intervention program.

CONTACTS AND LOCATIONS:
Locations (1):
- Nepal Health Research Council, Kathmandu, Bagmati, Nepal